CLINICAL TRIAL: NCT02908009
Title: An Observational Case Control Study to Identify the Role of Epigenetic Regulation of Genes Responsible for Energy Metabolism and Mitochondrial Function in the Obesity Paradox in Cardiac Surgery
Brief Title: A Case Control Study to Identify the Role of Epigenetic Regulation of Genes Responsible for Energy Metabolism and Mitochondrial Function in the Obesity Paradox in Cardiac Surgery
Acronym: Ob-Card
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0574
Record Dates: First submitted 2016-07-19; First posted 2016-09-20 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: C.Surgical Procedure; Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Atrial Biopsy: A 0.5cm x 0.5cm section of the right atrial wall is routinely excised to allow cannulation of the left atrium for connection to the cardiopulmonary bypass machine. This segment is routinely discarded. We propose to collect this specimen immediately after it has been discarded.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, single-centre case control comparison of expression of target genes responsible for energy utilisation, mitochondrial function and oxidative stress and levels of histone acetylation/ DNA methylation in obese and non-obese adult cardiac surgery patients. The study aims to test several inter-related hypotheses in a consecutive sequence of patients undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-existing paroxysmal, persistent or chronic atrial fibrillation,

Exclusion Criteria:

* Patients with pre-existing inflammatory state: sepsis undergoing treatment, acute kidney injury within 5 days, chronic inflammatory disease, congestive heart failure.
* Emergency or salvage procedure.
* Ejection fraction <30 %.
* Patient in a critical preoperative state (Kidney Disease: Improving Global Outcomes (KDIGO) Stage 3 AKI [20] or requiring inotropes, ventilation or intra-aortic balloon pump).
* Pregnancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be carried out at a large tertiary academic cardiac surgery unit in the UK; the University Hospitals of Leicester NHS Trust. This unit performs over 1,200 major cardiac procedures per year, of which 600 are patients undergoing coronary artery bypass grafting
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-09-09 (Actual); Primary Completion 2024-10-07 (Estimated); Study Completion 2024-10-07 (Estimated)

PRIMARY OUTCOMES:
Post surgery inotrope score | inotrope score measured up to 48 hours post-surgery
  inotrope score measured up to 48 hours post-surgery

SECONDARY OUTCOMES:
Changes in expression of target genes | Collected at the time of surgery
  from right atrial biopsies
Changes in epigenetic regulation of target genes from left atrial biopsies. | Collected at the time of surgery
  histone acetylation, DNA methylation
Changes in mitochondrial function | before and after sugery (up to 12 hours post surgery)
  in atrial biopsies and buffy coats of blood samples collected before and after surgery
Myocardial Injury | baseline and 24 hours
  defined by post cardiac surgery serum Troponin levels
Acute kidney injury | baseline, and up to 15 days post surgery (discharge)
  defined by serum creatinine level postoperatively, as per the KDIGO criteria
Perioperative clinical characteristics | Collected pre op
  Perioperative clinical characteristics
Perioperative medications. | Collected pre op
  Perioperative medications.
Data to calculate Multiple Organ Dysfunction (MOD) score. | baseline, and up to 96 hours post surgery
  To calculate the MOD score, the Respiratory Function (calculated as partial pressure of oxygen (PaO2) divided by fraction of inspired oxygen (FiO2)), Cardiovascular (Pressure adjusted heart rate (PAR) ), Renal (Serum Creatinine), Hepatic (serum bilirubi
Data to capture Acute Respiratory Distress Syndrome (Berlin criteria ARDS). | baseline, and up to 96 hours post surgery
  Acute Lung Injury (ALI) non-ARDS, ARDS. To define these different categories of acute lung injury, the Positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP) will be recorded in the CRF at time points: Pre-OP, ICU, 12 hrs post-op,24hrs post-op,48hrs post-op,72hrs post-op and 96hrs post-op. Along with the PaO2/FiO2 ratio, it will then be possible to categorise patients into the above definitions of acute lung injury as follows: ALI non-ARDS (200 mmHg <PaO2/FiO2<300 mmHg, regardless of PEEP),ARDS (PaO2/FiO2<200 mmHg, regardless of PEEP), mild Berlin Definition(200mmHg <PaO2/FiO2<300mmHg with PEEP > 5cm H2O),moderate Berlin Definition(100mmHg <calculated as partial pressure of oxygen divided by fraction of inspired oxygen PaO2/FiO2 < 200mmHg with PEEP > 5cm H2O) and Severe Berlin Definition (PaO2/FiO2 < 100mmHg with PEEP > 5cm H2O)
Data on demographics | Pre Op
  Height in cms
Data on demographics | Pre Op
  Weight in kgs

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Murphy, Principal Investigator — University of Leicester; Filiberto Serraino, Principal Investigator — University of Leicester
Locations (1):
- England, Glenfield, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Derived] Adebayo AS, Roman M, Zakkar M, Yusoff S, Gulston M, Joel-David L, Anthony B, Lai FY, Murgia A, Eagle-Hemming B, Sheikh S, Kumar T, Aujla H, Dott W, Griffin JL, Murphy GJ, Wozniak MJ. Gene and metabolite expression dependence on body mass index in human myocardium. Sci Rep. 2022 Jan 26;12(1):1425. doi: 10.1038/s41598-022-05562-8. PMID 35082386